CLINICAL TRIAL: NCT00099177
Title: A Randomized, Double-blind Study of the Effect of Bondronat Compared With Zoledronic Acid on Pain in Patients With Malignant Bone Disease Experiencing Moderate to Severe Pain
Brief Title: A Study to Assess the Efficacy of Intravenous/Oral Bondronat (Ibandronate) in Patients With Metastatic Bone Disease Experiencing Moderate to Severe Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO18039
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Pain; Bone Neoplasm; Neoplasm Metastasis
MeSH Terms: conditions — Pain; Bone Neoplasms; Neoplasm Metastasis | interventions — Ibandronic Acid; Zoledronic Acid

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bondronat]
- 2 (Active Comparator)
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: ibandronate [Bondronat] — 6mg iv on days 1-3, and 50mg po from day 22 to week 24
  Arms: 1
Drug: zoledronic acid — 4mg iv on day 1, and every 3-4 weeks
  Arms: 2

SUMMARY:
This 2 arm study will compare the efficacy of a regimen of intravenous (iv) and oral Bondronat with that of zoledronic acid in patients with malignant bone disease experiencing moderate to severe pain. Patients will be randomized to receive either Bondronat (6mg iv on days 1, 2 and 3 followed by Bondronat 5Omg po daily from day 22 to week 24) or zoledronic acid (4mg iv on day 1, and then every 3-4 weeks). The anticipated time of study treatment is 6-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients with malignant bone disease;
* patients with moderate to severe pain.

Exclusion Criteria:

* patients who have received a bisphosphonate within 3 weeks from the signing of informed consent;
* patients receiving concurrent investigational therapy, or who have received investigational therapy within 30 days of the first scheduled day of dosing;
* untreated esophagitis or gastric ulcers;
* recent or pre-scheduled radiotherapy to bone;
* patients who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain, as measured by Brief Pain Inventory and analgesic use | Week 24

SECONDARY OUTCOMES:
Performance score and QoL measures | Week 24
AEs and laboratory parameters | Throughout study
Opioid side effects | Throughout study
Skeletal-related events | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- United States (3):
  - Miami, Florida
  - Macon, Georgia
  - Houston, Texas
- Argentina (4):
  - Bahía Blanca
  - Buenos Aires
  - Rosario
  - Santa Fe
- Australia (2):
  - Adelaide
  - Brisbane
- Chile (2):
  - Santiago
  - Viña del Mar
- Hamburg, Germany
- Greece (2):
  - Kalyftaki Kifissia
  - Thessaloniki
- Guatemala City, Guatemala
- Hungary (3):
  - Budapest
  - Deszk
  - Szeged
- Italy (2):
  - Rozzano
  - Torino
- Mexico (4):
  - La Paz
  - Mexicali
  - Mexico City
  - Monterrey
- Panama City, Panama
- Poznan, Poland
- San Juan, Puerto Rico
- Russia (4):
  - Kazan'
  - Moscow
  - Obninsk
  - Saint Petersburg
- Sankt Gallen, Switzerland
- United Kingdom (2):
  - Manchester
  - Sutton